CLINICAL TRIAL: NCT07213648
Title: Modification of Threat Interpretation Bias to Reduce Anxiety in Neurodegenerative Movement Disorders (Aim 3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jessie Gibson, PhD, RN, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR 220251; K23NR020210 (NIH)
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Huntington Disease; Parkinson Disease
Keywords: CBM-I; cognitive bias modification; interpretation bias; anxiety; mobile app; Huntington; Parkinson
MeSH Terms: conditions — Huntington Disease; Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MindTrails-Movement CBM-I Condition (Experimental): The intervention group (N=68) will include participants with Huntington's disease (N=34) and Parkinson's disease (N=34). Participants will download the MindTrails-Movement app with active CBM-I training condition and will be prompted to complete brief, daily CBM-I training sessions for a period of 6 weeks. They will complete surveys assessing mood symptoms and interpretation bias at baseline, end of week 2, end of week 4, and end of week 6 (end of intervention), then again at the end of week 10.
  Interventions: Behavioral: MindTrails-Movement
- Waitlist Control Condition (Other): The waitlist control group (N=68) will include participants with Huntington's disease (N=34) and Parkinson's disease (N=34). Participants will be asked to download a control version of the app that includes access to a list of support resources but does not include daily CBM-I training content. They will complete surveys assessing mood symptoms and interpretation bias at baseline, end of week 2, end of week 4, and end of week 6, and end of week 10. Waitlist control participants will be offered the opportunity to complete the intervention version of the app after they complete their final study assessments.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: MindTrails-Movement — CBM-I training app with active CBM-I training condition
  Arms: MindTrails-Movement CBM-I Condition
Other: Waitlist Control — Version of MindTrails-Movement app including surveys and list of support resources but without active CBM-I training component
  Arms: Waitlist Control Condition

SUMMARY:
The purpose of this study is to assess preliminary efficacy of a tailored cognitive bias modification for interpretation (CBM-I) app for reducing anxiety in Huntington's disease and Parkinson's disease.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized controlled trial of the MindTrails-Movement CBM-I app in patients with Huntington's disease and Parkinson's disease (N=136). Participants randomly assigned to the intervention group (N=68) will be asked to download the MindTrails-Movement mobile app and to complete daily CBM-I training sessions and nightly surveys, in addition to surveys at baseline and every 2 weeks for the duration of the 6-week intervention and at 4-week follow-up (week 10).

Participants assigned to the waitlist control group will download a control version of the app without CBM-I training sessions. They will be asked to complete surveys in the app at baseline and every 2 weeks for the duration of the 6-week intervention and at 4-week follow-up (week 10). After 10 weeks, they will be offered the opportunity to access the version of MindTrails-Movement with CBM-I training content.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Huntington's disease or Parkinson's disease (genetic diagnosis of HD also acceptable)
* With anxiety symptoms (NeuroQoL Anxiety ≥12)

Exclusion Criteria:

* Cognitive decline precluding ability to consent or complete the intervention (MoCA 5 min/telephone ≤11)
* Unable to read and understand English
* Does not have regular access to an internet-connected device, capable of downloading and installing the mobile application (i.e., tablet or iPhone running iOS 10 or later or an Android phone running Android 5.0 or later)
* Not located in the USA
* <21 years old
* Active suicidality based on the answer "yes" to questions 4, 5, or 6b of the Columbia-Suicide Severity Rating Scale (Screen version)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Neurological Disorders (NeuroQoL) Anxiety short form | From baseline to end of week 6
  Patient-reported anxiety symptoms will be measured using the Quality of Life in Neurological Disorders Anxiety short form (NeuroQoL-Anxiety) total raw scores. This measure includes 8 items ranked 1-5, where the total score is the sum of item scores (range 8-40), and higher scores indicate worse anxiety symptoms.

SECONDARY OUTCOMES:
Movement Disorders Interpretation Bias Scale (MDIB) | From baseline to end of week 6
  Movement Disorders Interpretation Bias Scale (MDIB) is a measure of interpretation bias in people with movement disorders. Participants rate the likelihood (0-4) of three alternate explanations (two benign and one negative) for why an ambiguous event occurred. To obtain negative external and internal bias scores, the mean of 5 negative ratings for external threats (Items 3c, 5a, 7a, 10a, 11c) and the mean of 4 negative ratings for internal threats (Items 1b, 4c, 8b, 12b) will be computed, where higher scores (possible range: 0-4) reflect more severe negative interpretation biases.
Parkinson Anxiety Scale (PAS) | From baseline to end of week 6
  The Parkinson Anxiety Scale (PAS) total score will be used as a secondary measure of patient-reported anxiety symptoms. PAS includes 12 self-report items that make up three subscales (persistent and episodic anxiety and avoidant behavior). Items are ranked 0-4 with a maximum total score of 48, where higher scores indicate worse anxiety symptoms.
Brief Body Sensations Interpretation Questionnaire (BBSIQ) | From baseline to end of week 6
  Brief Body Sensations Interpretation Questionnaire (BBSIQ) is a general measure of interpretation bias. Participants rate the likelihood (0-4) of three alternate explanations (two benign and one negative) for why an ambiguous event occurred. To obtain negative external and internal bias scores, the mean of 7 negative ratings for external threats (Items 1c, 4c, 6a, 7b, 9b, 10b, 13c) and the mean of 7 negative ratings for internal threats (Items 2b, 3c, 5a, 8c, 11b, 12a, 14c) will be computed, where higher scores (possible range: 0-4) reflect more severe negative interpretation biases.

OTHER OUTCOMES:
Quality of Life in Neurological Disorders (NeuroQoL) Depression short form | From baseline to end of week 6
  Patient-reported depressive symptoms will be measured using the Quality of Life in Neurological Disorders Depression short form (NeuroQoL-Depression) total raw scores. This measure includes 8 items ranked 1-5, where the total score is the sum of item scores (range 8-40), and higher scores indicate worse depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Virginia School of Nursing, Charlottesville, Virginia, United States